CLINICAL TRIAL: NCT07098416
Title: An In-Depth Analysis of the Present Diagnostic and Therapeutic Landscape for Renal Anemia in China's Real-World Clinical Environment: A Multicenter Retrospective Cohort Investigation（DASHENG Study）
Brief Title: A Real-World Study About Anemia in Chronic Kidney Disease in China（DASHENG）
Acronym: DASHENG
Status: Not yet recruiting | Type: Observational
Sponsor: Wei Chen (Other)
Responsible Party: Sponsor-Investigator, Wei Chen, Doctor, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Other Study IDs: IIT-2025-121
Record Dates: First submitted 2025-07-10; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Anemia in Chronic Kidney Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Anemia affects the quality of life of CKD patients and increases the risk of CKD progression. we conducted a real-world study on patients with anemia in CKD to analyze the disease characteristics and treatment in Chinese patients with CKD-anemia.

DETAILED DESCRIPTION:
Anemia adversely affects the quality of life of CKD patients and increases the risk of CKD progression.

This study utilize data from approximately 20 medical centers across China. It aims to:

1. Analyze the disease characteristics, current diagnostic and treatments in Chinese patients with CKD-anemia.
2. Evaluate the safety and efficacy profiles of different drugs used for CKD-anemia.
3. Explore the direct medical costs associated with CKD-anemia management within real-world clinical practice in China.

ELIGIBILITY:
Inclusion Criteria: CKD patients will be defined as those meeting any of the following criteria during the observation period:

1. diagnosis of CKD (e.g., "%chronic kidney disease%", "%chronic nephropathy%", "%renal failure%", "%nephritis%" for complete ICD-9/10 code mapping*)
2. record of hemodialysis (HD) or peritoneal dialysis (PD) (refer to Attachment 2 for dialysis identification algorithms)
3. ≥2 eGFR measurements <60 mL/min/1.73m² (calculated using CKD-EPI equation) with ≥3-month interval (excluding acute kidney injury)

Exclusion Criteria:

1. Non-renal anemia due to trauma, traffic accidents, major hemorrhage, or other confirmed etiologies (e.g., acute hemorrhagic anemia, nutritional deficiency anemia, hemolytic anemia);
2. Diagnosis of acute kidney disease (AKD) without chronic kidney disease (CKD) comorbidity;
3. Incomplete critical data elements (including age, sex, or visit dates).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Anemia in Chronic Kidney Disease
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Disease characteristics and current treatments of anemia in chronic kidney disease (CKD) patients in China. | 20230101-20241231
  Disease characteristics and current treatments of anemia in chronic kidney disease (CKD) patients in China will beperformed to assess the proportions of CKD primary diseases, distribution of CKD stages, baseline Hb level distribution, and proportion of anti-anemia medication usage.
Incidence of Adverse Events according to CTCAE 5.0 (Safety profile of different anemia medications in CKD patients with anemia.) | 20230101-20241231
  An analysis will be performed to assess the safety according to CTCAE 5.0 .

SECONDARY OUTCOMES:
Analyze the efficacy of different anemia drugs in CKD patients with anemia. | 20230101-20241231
  Use the hemoglobin level to analyze the efficacy of different anemia drugs in CKD patients with anemia.
Explore the economic burden of anemia in CKD patients | 20230101-20241231
  Use the annual cost to explore the direct economic burden of anemia in CKD patients.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No